CLINICAL TRIAL: NCT04473261
Title: Efficacy of Iodine Complex in Mild to Moderate COVID-19 Patients
Brief Title: Efficacy of Iodine Complex Against COVID-19 Patients
Acronym: I-COVID-PK
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohaib Ashraf (Other)
Responsible Party: Sponsor-Investigator, Sohaib Ashraf, Post-Graduate Resident Cardiology, Sheikh Zayed Federal Postgraduate Medical Institute
Organization: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZMC/IRB/Internal/216/2020
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Covid19; SARS-CoV-2; Corona Virus Infection
Keywords: SARS-Cov-2; COVID-19; Coronavirus; Iodine Complex
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Capsules

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, multi-armed, close-label, interventional study designed
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: empty capsule will be given as a placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Iodine Complex (Capsule form) (Experimental): Iodine Complex) capsule (200mg) will be given three times a day
  Interventions: Drug: Iodine Complex
- Iodine Complex (Syrup form) (Experimental): Iodine Complex syrup form (40ml) will be given three times a day
  Interventions: Drug: Iodine Complex
- Standard Care Alone (Placebo Comparator): Placebo as empty capsule. Treatment will be given for all 4 arms will be receiving standard care as per version 3.0 of clinical management guidelines for COVID-19 established by the Ministry of National Health Services of Pakistan COVID-19 guidelines of the study setting.
  Interventions: Drug: Placebo
- Iodine Complex (Nasal Spray) (Experimental): Iodine complex throat spray of 2 puffs three times a day.
  Interventions: Drug: Idoine Complex

INTERVENTIONS:
Drug: Iodine Complex — Iodine Complex capsule (200mg) will be given three times a day
  Arms: Iodine Complex (Capsule form)
Drug: Iodine Complex — Iodine Complex syrup form (40ml) will be given three times a day
  Arms: Iodine Complex (Syrup form)
Drug: Placebo — Empty capsule will be given as placebo
  Other Names: capsule
  Arms: Standard Care Alone
Drug: Idoine Complex — Iodine Complex spray form 2 puffs will be given three times a day
  Arms: Iodine Complex (Nasal Spray)

SUMMARY:
The objective of this study is to measure the effect of Iodine complex in treating the COVID-19 patients to clear viral load of SARS-CoV-2 along with reduction in severity of symptoms and length of hospitalization of patients with COVID-19.

DETAILED DESCRIPTION:
The proposed study is a placebo-controlled, add-on, randomized trial using parallel group designs. This is a close-label and adaptive, multi-centered design with 1:1:1:1 allocation ratio and superiority framework.

ELIGIBILITY:
Inclusion Criteria:

* Positive PCR with mild to moderate disease

Exclusion Criteria:

* Allergic to iodine
* Any co-morbidity other than hypertension and dietetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
qRT-PCR | 14 days
  Time taken for viral load clearance
HRCT chest | 14 days
  Time taken for radiological improvement

SECONDARY OUTCOMES:
Severity of Symptoms | 14 days
  Time taken for symptomatic response in patients

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ashraf, PhD, Study Chair — University of Veterinary & Animal Sciences, Pakistan; Shoaib Ashraf, PhD, Study Director — Harvard University, Massachusetts General Hospital, Boston, USA; Moneeb Ashraf, MBBS, Principal Investigator — Mayo Hospital, Pakistan; Sohaib Ashraf, MBBS, Principal Investigator — Shaikh Zayed Medical Complex, Pakistan
Locations (1):
- Shaikh Zayed Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ashraf S, Ashraf S, Ashraf M, Farooq I, Akmal R, Imran MA, Kalsoom L, Ashraf S, Rafique S, Ghufran M, Akram MK, Sohaib-Ur-Rehman, Nadeem MF, Matti N, Siddiqui UN, Humayun A, Saboor QA, Ahmad A, Ashraf M, Izhar M; DOCTORS LOUNGE consortium. Clinical efficacy of iodine complex in SARS-CoV-2-infected patients with mild to moderate symptoms: study protocol for a randomized controlled trial. Trials. 2022 Jan 19;23(1):58. doi: 10.1186/s13063-021-05848-8. PMID 35045888
- [Derived] Ashraf S, Ashraf S, Ashraf M, Imran MA, Kalsoom L, Siddiqui UN, Farooq I, Ghufran M, Khokhar RA, Akram MK, Shahid I, Sohaib Ur Rehman M, Akmal R, Tahir A, Zahid A, Ashraf S, Rafique S, Matti N, Nadeem MF, Humayun A, Malik A, Saboor QA, Ahmad A, Ashraf M, Izhar M. A quadruple blinded placebo controlled randomised trial to evaluate the effectiveness of an Iodine complex for patients with mild to moderate COVID-19 in Pakistan (I-COVID-PK): A structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Feb 10;22(1):127. doi: 10.1186/s13063-021-05081-3. PMID 33568226